CLINICAL TRIAL: NCT03109678
Title: A Comparison of the Intubating Laryngeal Mask FASTRACH™ and the Intubating Laryngeal Mask Ambu Aura-i™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asklepios Kliniken Hamburg GmbH (Other)
Collaborators: University of Kiel (Other)
Responsible Party: Principal Investigator, Dr. Robert Schiewe, Doctor, Asklepios Kliniken Hamburg GmbH
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: AZ 107/02
Record Dates: First submitted 2017-03-08; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Airway Management; Laryngeal Mask Airway; Fibreoptic Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aura-i / Rüsch (Experimental): Blind tracheal intubation: Combination of laryngeal mask Ambu Aura-i™ with Rüsch Super Safety Silk™ tracheal tube
  Interventions: Device: Crossover Ambu Aura-i™ / Rüsch Super Safety Silk™
- Aura-i / LMA ETT (Experimental): Blind tracheal intubation: Combination of laryngeal mask Ambu Aura-i™ with LMA ETT™ tracheal tube
  Interventions: Device: Crossover Ambu Aura-i™ / LMA ETT™
- Fastrach / Rüsch (Experimental): Blind tracheal intubation: Combination of laryngeal mask Fastrach™ with Rüsch Super Safety Silk™ tracheal tube
  Interventions: Device: Crossover FASTRACH™ / Rüsch Super Safety Silk™
- Fastrach / LMA ETT (Experimental): Blind tracheal intubation: Combination of laryngeal mask Fastrach™ with LMA ETT™ tracheal tube
  Interventions: Device: Crossover FASTRACH™ / LMA ETT™

INTERVENTIONS:
Device: Crossover Ambu Aura-i™ / Rüsch Super Safety Silk™ — After unsuccessful blind intubation in the Ambu Aura-i™ / Rüsch Super Safety Silk™ group: crossover design using the Ambu Aura-i™ mask in combination with the LMA ETT™ tracheal tube
  Arms: Aura-i / Rüsch
Device: Crossover Ambu Aura-i™ / LMA ETT™ — After unsuccessful blind intubation in the Ambu Aura-i™ / LMA ETT group: crossover design using the Ambu Aura-i™ mask in combination with the Rüsch Super Safety Silk™ tracheal tube
  Arms: Aura-i / LMA ETT
Device: Crossover FASTRACH™ / Rüsch Super Safety Silk™ — After unsuccessful blind intubation in the FASTRACH™ / Rüsch Super Safety Silk™ group: crossover design using the FASTRACH™ mask in combination with the LMA ETT™ tube
  Arms: Fastrach / Rüsch
Device: Crossover FASTRACH™ / LMA ETT™ — After unsuccessful blind intubation in the FASTRACH™ / LMA ETT™ group: crossover design using the FASTRACH™ mask in combination with the Rüsch Super Safety Silk™ tube
  Arms: Fastrach / LMA ETT

SUMMARY:
The intubating laryngeal mask Fastrach™ is considered a gold standard for blind intubation as well as for fibreoptic guided intubation via a laryngeal mask. Recently, a single use version of the mask has been introduced. The Fastrach single use laryngeal mask is beng compared to the new, low-priced single use intubating laryngeal mask Ambu Aura-i™.

DETAILED DESCRIPTION:
Eighty patients undergoing general anaesthesia with planned tracheal intubation for elective surgical procedures are enrolled in the study after checking for inclusion and exclusion criteria. Patients are randomised to either LMA group for blind tracheal intubation with either a standard PVC tracheal tube, or a specifically for the LMA Fastrach developed tube, yielding 4 subgroups.

After a standardised anaesthesia induction, blind intubation is performed in each study group. Different time intervals are documented, such as time to first adequate lung ventilation, or f.e. time for laryngeal mask placement. A crossover-design is performed after unsuccessful intubation, using the alternate LMA or the other tracheal tube. LMA placement is visualised by fibreoptic control.

An estimated success rate for blind intubation of 60% in the Aura-i group versus 90% in the Fastrach group yields a sample size of n= 38. To compensate for dropouts, n=40 subjects are enrolled in each group.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing planned general anaesthesia
* planned tracheal intubation
* elective surgical procedure
* 15 to 80 years of age

Exclusion Criteria:

* ASA physical status IV and V
* severe pulmonary comorbidity (COPD GOLD >III, bronchial asthma)
* indication for rapid-sequence induction
* mouth opening (interincisor distance) <3cm
* morbid obesity (BMI >35kg.m-2)

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-07-12 (Actual); Primary Completion 2012-03-07 (Actual); Study Completion 2012-03-07 (Actual)

PRIMARY OUTCOMES:
success rate of blind intubation | through study completion; time frame for individual study patient: two attempts of blind tracheal intubation peri-interventional, time maximum of 300 seconds
  overall success rate of blind tracheal intubation within two attempts using either the FASTRACH™ laryngeal mask or the Ambu Aura-i™ laryngeal mask

SECONDARY OUTCOMES:
influence of tracheal tubes | through study completion; time frame for individual study patient: two attempts of blind tracheal intubation peri-interventional, time maximum of 300 seconds
  influence of success rates of blind tracheal intubation using different tracheal tubes (Rüsch or LMA-ETT)
equivalence of the laryngeal masks regarding fibreoptic visualisation | through study completion; after placing the laryngeal mask and checking for airway leak pressure, fibreoptic visualisation is performed within 60 seconds
  fibreoptic control of laryngeal mask placement (Fastrach and Aura-i); the position of the larynx relative to the laryngeal cuff and mask-aperture is visualised and categorised as "correct", "lateral deviation", "epiglottic downfolding" or "not assessable"; additionally, the view on the larynx comparable to Cormack/Lehane score is recorded
subjective handling score | through study completion; the handling of the laryngeal masks during the first placement attempt within 60 seconds; directly after placing laryngeal masks and before fibreoptic visualisation, the subjective handling score is documented as above
  subjective handling score for the two compared laryngeal masks, rated as excellent (1) - poor (4)
differences in airway leak pressure | through study completion; right after placing the laryngeal mask and checking for correct positioning, ALP is documented within 60 seconds
  differences in airway leak pressure (ALP) of the two compared laryngeal masks, in cm H2O; presence of audible leakage as well as the absence of corresponding pressure increase on the monitor recorded by setting the APL valve to 40cm H2O, and fresh gas flow at 3l/min
incidence of postoperative sore throat and hoarseness | patient interview 24 hours post procedural
  incidence of postoperative sore throat and hoarseness as well as difficulty swallowing as reported by the study patients ("none", "moderate", "severe")

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Bein, Prof. Dr., Study Chair — Asklepios Kliniken Hamburg GmbH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schiewe R, Stoeck M, Gruenewald M, Hoecker J, Bein B. A comparison of blind intubation with the intubating laryngeal mask FASTRACH and the intubating laryngeal mask Ambu Aura-i a prospective randomised clinical trial. BMC Anesthesiol. 2019 Mar 30;19(1):44. doi: 10.1186/s12871-019-0718-6. PMID 30927922